CLINICAL TRIAL: NCT02662322
Title: Effect of Language and Confusion on Pain During Peripheral Intravenous
Brief Title: Effect of Language and Confusion on Pain During Peripheral Intravenous Catheterization (KTHYPE)
Acronym: KTHYPE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 35RC15_9868
Record Dates: First submitted 2016-01-12; First posted 2016-01-25 (Estimated); Last update posted 2018-05-07 (Actual); Status verified 2018-05

CONDITIONS: Anaesthesia
Keywords: Communication; Confusion; Intravenous Catheterization; Comfort
MeSH Terms: conditions — Communication; Confusion

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- HYPNOSIS (Experimental): hypnotic communication, confusion procedure during peripheral intravenous catheterization
  Interventions: Other: Hypnotic communication; Other: peripheral intravenous catheterization
- NOCEBO (Active Comparator): negative connotation communication during peripheral intravenous catheterization
  Interventions: Other: negative connotation communication; Other: peripheral intravenous catheterization
- NEUTRAL (Placebo Comparator): neutral connotation communication during peripheral intravenous catheterization
  Interventions: Other: neutral connotation communication; Other: peripheral intravenous catheterization

INTERVENTIONS:
Other: Hypnotic communication — hypnotic communication during peripheral intravenous catheterization
  Arms: HYPNOSIS
Other: negative connotation communication — negative connotation communication during peripheral intravenous catheterization
  Arms: NOCEBO
Other: neutral connotation communication — neutral connotation communication during peripheral intravenous catheterization
  Arms: NEUTRAL
Other: peripheral intravenous catheterization — peripheral intravenous catheterization

SUMMARY:
The purpose of this study is to compare three communications during peripheral intravenous catheterization and measure pain patient: one hypnotic, confusion (HYPNOSIS), an other with negative connotation (NOCEBO) and at least with neutral connotation (NEUTRAL).

DETAILED DESCRIPTION:
Clinicians used to warn patients of pain or discomfort before potentially painful procedures like peripherical intravenous catheterization (PIVC). However, suggestions for negative perceptual experiences causes more pain and anxiety. During This does not improve at all the real-life experience of the act. On the contrary, the use of gentler words improves pain perception and subjective patient experience. Furthermore, hypnosis has been demonstrated as efficient and the pain perception seems to be modulate by hypnotic suggestions.

ELIGIBILITY:
Inclusion Criteria:

* at least 18 years
* peripheral intravenous catheterization of 20 G on the dorsal face of the hand before a planned surgery
* written and informed patient consent

Non inclusion Criteria:

* patient unable to communicate in french
* difficult vein access characteristics
* premedication
* pregnant, breast-feeding woman
* patient subject of legal protection

Exclusion criteria :

* failed of the first attempt of peripheral intravenous catheterization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 294 (Actual)
Dates: Start 2016-03-10 (Actual); Primary Completion 2017-03-06 (Actual); Study Completion 2017-09-06 (Actual)

PRIMARY OUTCOMES:
numerical rating scale for pain from 0 to 10 | data collected within 3 min after the end of peripheral intravenous catheterization procedure
  self-evaluation of pain catheterization

SECONDARY OUTCOMES:
evolution of numerical rating scale for comfort from 0 to 10 | data collected just before and within 3 min after peripheral intravenous catheterization procedure
  self-evaluation of comfort catheterization
evolution of numerical rating scale for anxiety from 0 to 10 | data collected just before and within 3 min after peripheral intravenous catheterization procedure
  self-evaluation of anxiety catheterization
presence of spontaneous patient arm withdrawal | data collected within 3 min after the end of peripheral intravenous catheterization procedure
presence of unprompted vocalization by word(s) or sound(s) | data collected within 3 min after the end of peripheral intravenous catheterization procedure

CONTACTS AND LOCATIONS:
Overall Officials: Helene Beloeil, PH, Principal Investigator — Rennes University Hospital
Locations (3):
- Cliniques Universitaires Saint-Luc, Brussels, Belgium
- France (2):
  - CHU, Rennes
  - Centre Hospitalier Privé Saint Grégoire, Saint-Grégoire

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fusco N, Bernard F, Roelants F, Watremez C, Musellec H, Laviolle B, Beloeil H; Effect of Language and Confusion on Pain During Peripheral Intravenous Catheterization (KTHYPE) group. Hypnosis and communication reduce pain and anxiety in peripheral intravenous cannulation: Effect of Language and Confusion on Pain During Peripheral Intravenous Catheterization (KTHYPE), a multicentre randomised trial. Br J Anaesth. 2020 Mar;124(3):292-298. doi: 10.1016/j.bja.2019.11.020. Epub 2019 Dec 18. PMID 31862159